CLINICAL TRIAL: NCT00863629
Title: Tight Glycemic Control Increases Cardiac Stem Cells and Reduces Heart Remodeling During Acute Myocardial Infarction in Hyperglycemic Patients
Brief Title: Tight Glycemic Control Increases Cardiac Stem Cells During Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Raffaele Marfella, MD, PhD, Second University of Naples, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-4546789
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Myocardial Infarction; Oxidative Stress; Glycemic Control
Keywords: myocardial infarction; oxidative stress; stem cells; glycemic control
MeSH Terms: conditions — Myocardial Infarction | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): 25 normoglycemic patients as control group
- 2 (Active Comparator): 20 hyperglycemic patients (glucose >140 mg/dl) randomized to conventional glycemic control by insulin (CGC group; glucose goal 180-200 mg/dl)
  Interventions: Drug: Insulin
- 3 (Experimental): 20 hyperglycemic patients (glucose >140 mg/dl) were randomized to intensive glycemic control by insunin (IGC group; glucose goal 80-140 mg/dl)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — In the CGC group, continuous insulin infusion was started only when blood glucose levels exceeded 200 mg/dl and adjusted to keep blood glucose between 180 and 200 mg/dl. When blood glucose fell <180 mg/dl, insulin infusion was tapered slowed down and eventually stopped. In the IGC group, insulin infusion was started when blood glucose levels exceeded 140 mg/dl and adjusted to maintain glycemia at 80-140 mg/dl. After the start of insulin infusion protocol a glycemic control was provided every hour in order to obtain three consecutive values that were within the goal range. Plasma glucose levels were checked every two hours in both CGC and IGT patients throughout the study period. The infusion lasted until stable glycemic goal (ICG group: 80-140 mg/dl; CGC group: 180-200 mg/dl) at least for 24 h. Subcutaneous insulin was initiated at the cessation of the infusion. Insulin was given as short-acting insulin before meals and intermediate long-acting insulin in the evening, in both group.
  Arms: 2; 3

SUMMARY:
Objectives. The investigators analysed the effects of tight glycemic control in regenerative potential of the myocardium during acute myocardial infarction (AMI).

Background. A strict glycemic control after AMI improves the cardiac outcome. The role of tight glycemic control in regenerative potential of the myocardium during acute myocardial ischemia are still largely unknown.

Methods. Sixty-five patients with first AMI undergoing coronary bypass surgery were studied: 25 normoglycemic patients served as control group; hyperglycemic patients (glucose >140 mg/dl) were randomized to intensive glycemic control (IGC, n=20; glucose goal 80-140 mg/dl) or conventional glycemic control (CGC, n=20; glucose goal180-200 mg/dl) for almost 3 days before surgery, using insulin infusion followed by subcutaneous insulin treatment. Echocardiographic parameters were investigated at admission and after treatment period. During surgery, oxidative stress (nitrotyrosine, O2- production), apoptosis (Caspase-3) and cardiac stem cells (CSCs) (c-kit, MDR1 and Sca-1 positive cells) were analysed in biopsy specimens taken from the peri-infarcted area.

DETAILED DESCRIPTION:
The study design was structured on the basis of protocol Yale . Upon emergency wards admission, hyperglycemic patients were randomly assigned to IGC or CGC. In patients with STEMI the insulin infusion was started after thrombolysis. In the CGC group, continuous insulin infusion of 50 IU Actrapid HM (Novo Nordisk) in 50 ml NaCl (0.9% using a Perfusor-FM pump) was started only when blood glucose levels exceeded 200 mg/dl and adjusted to keep blood glucose between 180 and 200 mg/dl. When blood glucose fell <180 mg/dl, insulin infusion was slowed down and eventually stopped. In the IGC group, insulin infusion was started when blood glucose levels exceeded 140 mg/dl and adjusted to maintain glycemia at 80-140 mg/dl. During insulin infusion, oral feeding was stopped and parenteral nutrition (13±5 Kcal/kg-1/day-1) was started. After the start of insulin infusion protocol a glycemic control was provided every hour in order to obtain three consecutive values that were within the goal range. Capillary glucose levels were measured by fingerstick testing. Additionally, plasma glucose levels were checked every two hours in both CGC and IGT patients throughout the study period. Both measurements were no statistically different . The infusion lasted until stable glycemic goal (ICG group: 80-140 mg/dl; CGC group: 180-200 mg/dl) at least for 24 h. After glycemic goal were maintained for 24 h, a parenteral nutrition was stopped and feeding was started according to European guidelines (10). Subcutaneous insulin was initiated at the cessation of the infusion. Insulin was given as short-acting insulin before meals and intermediate long-acting insulin in the evening, in both group. In IGC group, the treatment goal was a fasting blood glucose level of 90-140 mg/dl and a non-fasting (two hours after meal) level of <180 mg/dl (4). In CGC group, the treatment goal was fasting blood glucose and postprandial levels of <200 mg/dl. With regard to the full medical therapy, the protocol stated that the use of concomitant treatment should be as uniform as possible and according to evidence-based international guidelines for AMI.

Echocardiographic assessment. Patients enrolled in the study underwent two-dimensional echocardiography at admission before starting full medical therapy as well as after achieved glycemic control goal for almost 3 days, before surgery. The study was performed using a standardized protocol and phased-array echocardiographs with M-mode, two-dimensional, and pulsed, continuous-wave, and color flow Doppler capabilities. The ejection fraction was calculated from area measurements using the area-length method applied to the average apical area. The left ventricular internal dimension and interventricular septal were measured at the end diastole and end systole, and the wall motion score index was calculated according to American Society of Echocardiography recommendations. Isovolumetric relaxation time (IRT) was the time interval from cessation of left ventricular outflow to onset of mitral inflow, the ejection time (ET) was the time interval between the onset and the cessation of left ventricular outflow, and the mitral early diastolic flow deceleration time was the time interval between the peak early diastolic flow velocity and the end of the early diastolic flow. The total systolic time interval was measured from the cessation of one mitral flow to the beginning of the following mitral inflow. Isovolumetric contracting time (ICT) was calculated by subtracting ET and IRT from the total systolic time interval. The ratio of velocity time intervals (vti) of mitral early (E) and late (A) diastolic flows (Evti/Avti) was calculated. The myocardial performance index (MPI) was calculated as (IRT+ICT)/ET.

Biopsy of myocardium. All patients were undergone to CABG after maintained glucose goal for almost 3 days. After induction of anaesthesia and median sternotomy, the heart of each patient was examined, and 3-mm partial-thickness biopsy specimens were taken from the peri-infarcted area. The infarcted zone was identified as a yellow area surrounded by a purple band of granulation tissue or as gray area with fine yellow lines at its periphery. The peri-infarct zone was identified as a zone immediately adjacent the zone with the anatomical characteristics of myocardial infarct. Moreover, the transesophageal echocardiogram (TEE) was performer to evaluate peri-infarct zone All biopsies were performed before CABG, during ventilation with a fraction of inspired oxygen of 40% and peripheral oxygen saturations of >95%.

Analysis of specimens. Half of each biopsy specimen was fixed in formalin, sectioned to a thickness of 5 µm, mounted on slides, and stained with hematoxylin and eosin. The mounted specimens were then examined for evidence of ischemia or kept for immunohistechemistry. The other half of the specimen was frozen in liquid nitrogen for Western Blotting analysis.

ELIGIBILITY:
Inclusion Criteria:

* evidence of AMI within the last 8 h (troponin-I >2.50 µg/l together with either typical symptoms of angina or electrographic criteria of ST-segment modification)
* first uncomplicated AMI
* the need for CABG

Exclusion Criteria:

* previous AMI
* inflammatory disorders
* malignancy
* renal diseases infections

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2001-01; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
cardiac stem cells during acute myocardial infarction | 3 days of treatment

SECONDARY OUTCOMES:
heart remodeling during acute myocardial infarction | 3 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Marfella, MD, PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Second University of Naples, Naples, Italy

REFERENCES:
- [Background] Kunz GA, Liang G, Cuculi F, Gregg D, Vata KC, Shaw LK, Goldschmidt-Clermont PJ, Dong C, Taylor DA, Peterson ED. Circulating endothelial progenitor cells predict coronary artery disease severity. Am Heart J. 2006 Jul;152(1):190-5. doi: 10.1016/j.ahj.2006.02.001. PMID 16824855
- [Background] Assmus B, Walter DH, Lehmann R, Honold J, Martin H, Dimmeler S, Zeiher AM, Schachinger V. Intracoronary infusion of progenitor cells is not associated with aggravated restenosis development or atherosclerotic disease progression in patients with acute myocardial infarction. Eur Heart J. 2006 Dec;27(24):2989-95. doi: 10.1093/eurheartj/ehl235. Epub 2006 Oct 19. PMID 17053006
- [Background] Pal R. Embryonic stem (ES) cell-derived cardiomyocytes: a good candidate for cell therapy applications. Cell Biol Int. 2009 Mar;33(3):325-36. doi: 10.1016/j.cellbi.2008.12.001. Epub 2008 Dec 14. PMID 19121644
- [Derived] Marfella R, Sasso FC, Cacciapuoti F, Portoghese M, Rizzo MR, Siniscalchi M, Carbonara O, Ferraraccio F, Torella M, Petrella A, Balestrieri ML, Stiuso P, Nappi G, Paolisso G. Tight glycemic control may increase regenerative potential of myocardium during acute infarction. J Clin Endocrinol Metab. 2012 Mar;97(3):933-42. doi: 10.1210/jc.2011-2037. Epub 2011 Dec 14. PMID 22170713